CLINICAL TRIAL: NCT02249533
Title: Evaluation of Spot Light: A Concussion Injury Management App for Youth Sports
Acronym: SpotLight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lara McKenzie (Other)
Responsible Party: Sponsor-Investigator, Lara McKenzie, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HD080377
Record Dates: First submitted 2014-01-29; First posted 2014-09-25 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: TBI
Keywords: Spot Light; High School RIO; Concussion; Injury Prevention; Football; Pop Warner; High School; Middle School
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spot Light and High School RIO (Experimental): A total of 200 youth football teams (100 high school and 100 middle school-aged teams) will be enrolled. Potential participating teams, all high schools eligible to report football data to High School RIO™ as well as all Pop Warner and Middle School sponsored football teams that have a valid e-mail contact, will be e-mailed a letter inviting them to participate (Appendix 3).
  Intervention: Certified Athletic Trainers will be given access to report football injuries via High School RIO and will report potential concussions using the Spot Light Concussion app.
  Interventions: Other: Spot Light Concussion App
- Control (No Intervention): Control: Certified Athletic Trainers will be given access to report football injuries via High School RIO.

INTERVENTIONS:
Other: Spot Light Concussion App — Certified Athletic Trainers will report football injuries using High School RIO and will report possible concussions using the Spot Light concussion app.
  Arms: Spot Light and High School RIO

SUMMARY:
Sports-related traumatic brain injuries (TBIs), including mTBIs-commonly referred to as concussions-are a serious public health concern. Diagnostic criteria and consensus return to play (RTP) guidelines exist, but clinicians have varying approaches to the diagnosis and management of sports-related concussion as these guidelines are almost completely unsupported by an evidence base. It is well known that by increasing awareness of concussion signs and symptoms as well as the importance of addressing this injury, improving coaching on proper sports activity techniques and good sportsmanship, providing appropriate protective equipment, and quickly responding to injuries, the incidence, severity, and long-term negative health effects of sports-related concussion among children and adolescents can be reduced. The overall objective of this application, which is the first step toward attainment of our long-term goal, is to evaluate the effectiveness of Spot Light (a concussion injury management application [app] that coordinates diagnosis, management, and RTP procedures from injury to safe return to sport) when utilized by youth football teams. Our central hypothesis is that youth football teams randomized to receive SpotLight will report increased rates of concussion, increased referrals to physicians for care, and increased athlete compliance with RTP guidelines. The rationale that underlies the proposed research is that providing an easy to-use app has a high probability of effectively helping people involved with youth sports better recognize, respond to, and ensure athletes are fully recovered from sports-related concussion. We will test our hypothesis by pursuing the following aims: 1: Evaluate whether Spot Light will increase reported rates of sports-related concussion; Aim 2: Evaluate whether Spot Light increases referrals to physicians following concussion; Aim 3: Evaluate whether Spot Light improves the management of sports-related concussion. We expect to determine whether there is increased reporting, referrals to physicians, and athlete compliance with RTP guidelines. This contribution will be significant because it will allow physicians, athletic trainers (ATs), coaches, and parents to collaboratively track concussions from injury through safe RTP thereby lessening the chances of long-term negative outcomes as well as acute catastrophic outcomes.

DETAILED DESCRIPTION:
Sports-related traumatic brain injuries (TBIs), including mTBIs - commonly referred to as concussions - are a serious public health concern. During the last decade, emergency department visits for sports and recreation related TBIs among youth, including concussions, increased by 62%.[1] Concussion rates among high school athletes have significantly increased over the past decade.[2] Although most sports-related concussions are mild injuries where the athlete fully recovers from symptoms within a week, [3-5] each year TBIs contribute to a substantial number of deaths and cases of permanent disability. While contact sports such as football have the highest incidence and rates of concussion, these injuries occur across a wide range of sports.[5] Diagnostic criteria and consensus return to play (RTP) guidelines exist, but clinicians have varying approaches to the diagnosis and management of sports-related concussions as these guidelines are almost completely unsupported by an evidence base. Increasing awareness of concussion signs and symptoms, improving sport specific coaching techniques, promoting good sportsmanship, providing appropriate protective equipment and responding quickly to injuries reduces the incidence, severity and long-term negative health effects of sports related concussions among children and adolescents.[1] Thus there is a critical need for the development of tools for prevention. Our long-term goal is to reduce the negative consequences of sports-related concussions, specifically in youth sports. The overall objective of this application, which is the first step toward attainment of our long-term goal, is to evaluate the effectiveness of Spot Light (a concussion injury management application [app] that organizes and coordinates diagnosis, management, and RTP procedures from injury to safe return to sport) (Appendix 1) when utilized by middle and high school football teams. Our central hypothesis is that middle and high school football teams randomized to receive Spot Light will report increased rates of concussion; increased referrals to physicians for care, and increased athlete compliance with RTP guidelines. The rationale that underlies the proposed research is that providing an easy-to-use app for sports-related concussions has a high probability of effectively helping people involved with youth sports better recognize, respond to, and ensure that athletes are fully recovered from sports-related concussion.

We plan to test our central hypothesis and, thereby, attain the objective of this application by pursuing the following specific aims: Aim 1. Evaluate whether or not Spot Light increases reported rates of sports-related concussions.

Working Hypothesis-teams using Spot Light will report a higher rate of concussion than teams without Spot Light.

Aim 2. Evaluate whether or not Spot Light increases referrals to physicians for patient care following a sports-related concussion. Working Hypothesis-teams using Spot Light will refer more concussed athletes for treatment by a physician than teams without Spot Light.

Aim 3. Evaluate whether or not Spot Light improves management of sports-related concussions.

Working Hypothesis-injured athletes on teams utilizing Spot Light will exhibit higher compliance with RTP guidelines, than teams without Spot Light.

It is anticipated that these aims will yield the following expected outcomes. We expect to determine whether there is increased reporting of concussion, referrals to physicians, and athlete compliance with RTP guidelines. We also expect to learn whether the app is adopted and utilized similarly when distributed to different levels of youth sports (middle vs. high school age) and different types of "reporters" (coaches vs. certified athletic trainers). We expect widespread effectiveness across age groups and types of reporters; these results would suggest that Spot Light is suitable for widespread distribution across a variety of youth sports and settings. These outcomes are expected to have an important positive impact because timely and proper diagnosis, management, and coordination of care and RTP decisions will ultimately reduce the negative consequences and impact of sports-related concussions, as will now be detailed in the next section.

ELIGIBILITY:
Inclusion Criteria:

* middle school or high school aged athletes
* "reporter" must have an iOS device, such as an iPhone, iPad, etc., and a valid email address
* reporter must be comfortable answering questions in English
* reporter must be willing to utilize the RIO™ system weekly throughout the season
* reporter must be willing to download the Spot Light app if randomized into the IG

Exclusion Criteria:

* already currently enrolled in the study under a different condition

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 175 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Central Hypothesis/Study Aim 1: Rates of Reported Concussions | 1 year (football season)
  Our central hypothesis is that middle and high school football teams randomized to receive Spot Light will report increased rates of concussion; increased referrals to physicians for care, and increased athlete compliance with RTP guidelines. We will compare the rates of concussions entered in the RIO system with those entered into the SpotLight Concussion Management System. Concussion rates are calculated by dividing concussion incidence (numerator) by athlete exposures (denominator). Any reportable concussion is one that: occurred as a result of an organized practice or competition during the past week whether or not it resulted in restriction of the athlete's participation. We will compare the intervention and control in terms of the reported concussion rate and the referred concussion events rate per 1,000 athlete-exposures from each team.

SECONDARY OUTCOMES:
Specific Aim 2: Physician Referrals | 1 year (football season)
  Aim 2. Evaluate whether or not Spot Light increases referrals to physicians for patient care following a sports-related concussion. We will examine the differences in the number of those referred to physician for follow-up care (yes/no) between our control and intervention group. We will compare the intervention and control in terms of the reported concussion rate and the referred concussion events rate per 1,000 athlete-exposures from each team.
Specific Aim 3: Management of Concussions | 1 year (football season)
  Aim 3. Evaluate whether or not Spot Light improves management of sports-related concussions. Data analytic activities for the proposed project will primarily be comprised of two activities: (1) the generation of descriptive information summarizing the sample and its characteristics; and (2) the analyses related to the aims and hypotheses. We will compare the intervention and control on demographic characteristics and other covariates using chi-square tests for categorical variable comparisons and t-tests for continuous variables as a check of the randomization. We will compare the intervention and control in terms of the reported concussion rate and the referred concussion events rate per 1,000 athlete-exposures from each team and the rate of complied events from each team. The number of athletes on each team, and the number of practices and competitions will be considered as covariates in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lara B McKenzie, PhD, Principal Investigator — Center for Injury Research and Policy The Research Insititute at Nationwide Children's Hospital
Locations (1):
- Center for Injury Research and Policy, Nationwide Children's Hospital, Columbus, Ohio, United States